CLINICAL TRIAL: NCT03897062
Title: A Placebo-controlled, Double -Blind Randomised Trial of Suvorexant in the Management Comorbid Sleep Disorder and Alcohol Dependence
Brief Title: Suvorexant in the Management Comorbid Sleep Disorder and Alcohol Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems during covid lockdowns resulted in Merck ceasing supply of suvorexant/placebo
Sponsor: The Florey Institute of Neuroscience and Mental Health (Other)
Collaborators: St Vincent's Hospital Melbourne (Other); Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49730
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Insomnia; Alcohol Use Disorder
Keywords: suvorexant; insomnia; alcohol use disorder; craving; withdrawal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcoholism | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: A placebo-controlled, double-blind randomised trial
Who Masked: Outcomes Assessor
Masking Description: Patients will be treated from pre-packaged blinded treatment schedules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Active Comparator): Patients (n=64): 20mg tablets of suvorexant nocte daily for six months
  Interventions: Drug: Suvorexant 20 mg
- Placebo group (Placebo Comparator): Placebo control group: Patients (n=64): 1 placebo tablet nocte daily for six months in addition to treatment as usual
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Suvorexant 20 mg — Placebo controlled double blind suvorexant vs placebo
  Arms: Treatment group
Other: placebo — Placebo controlled double blind suvorexant vs placebo
  Arms: Placebo group

SUMMARY:
Suvorexant (trade name Belsomra) is an orexin receptor antagonist that has TGA approval for the treatment of insomnia, characterised by difficulties with sleep onset and/or sleep maintenance. It may also have a role in addictions as the orexins play a critical role in drug addiction and reward-related behaviours. Orexins appear to be involved in both alcohol withdrawal and in alcohol seeking triggered by external cues (eg contexts or stressors) through both OX1 and OX2 receptor signalling. Chief investigator, Professor Lawrence was the first to demonstrate a role for endogenous orexin signaling in alcohol-seeking. Alcohol is known to effect the sleep of healthy and alcohol dependent individuals with effects on daytime sleepiness, physiological functions during sleep, and the development of sleep disorders. There are various estimates of the co-occurrence of insomnia and alcohol use disorder ranging from 36-72%. In alcohol dependent individuals sleep is disturbed both while drinking and for months of abstinence and abstinent sleep disturbance is predictive of relapse.

This proposal aims to evaluate the use of suvorexant as a safe and effective pharmacotherapy to treat sleep disorders in alcohol dependent patients undergoing acute alcohol withdrawal and thereafter for six months. The study will also examine the effectiveness of suvorexant in reducing craving for alcohol and promoting duration of abstinence. This will be the first double blind controlled trial of suvorexant in the management of the alcohol withdrawal syndrome and maintenance of abstinence post withdrawal.

DETAILED DESCRIPTION:
Study Procedures Baseline On Day 1, prior to commencement of treatment baseline data will be collected on demographics, ISI questionnaire plus 2 short questions 1) how many hours sleep has the participant had for the past week; 2) how would the participant rate their sleep quality in the past week. The investigators will also determine previous drug use history, physical examination, urine drug screen and measures of alcohol dependence severity, psychological and social functioning (ATOPv7).

Treatment Period Treatment will begin immediately after collection of Baseline data. Suvorexant will not be given if breath alcohol concentration is above zero. Both groups will be treated using the St Vincent's Hospital standard protocol for management of alcohol withdrawal, in which benzodiazepines are provided as required according to the symptoms listed in the Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar). That is, if the CIWA-Ar score is > 10 then benzodiazepines (BZD) are administered. Note, BZD will not be given for management of insomnia. Physicians involved in patient care, nurses and participants will be blinded to treatment assignment. Participants will be monitored for signs of adverse events (i.e. distress, significant alcohol withdrawal, and adverse response to suvorexant) approximately 4 hourly for the first 24 - 48 hrs of residential stay and then according to clinical assessment. All clinical observations will be made by a suitably qualified and experienced medical professional. Where any adverse events are observed, monitoring will be increased to meet clinical needs and treatment discontinued if required. Alcohol withdrawal severity will be assessed using the Clinical Institute Withdrawal Assessment - Alcohol revised (CIWA-Ar).

Note, during in-patient assessment there will be no consumption of alcohol (7-10 days). Upon release to outpatients the investigators will advise participants not to consume alcohol and will provide follow-up support to help maintain abstinence. If patients resume heavy drinking and are deemed to have relapsed i.e. daily alcohol consumption greater than 5 standard drinks each day, the investigators will tell them to cease the medication and they will be withdrawn from the study. Data collected to this point will be included in the study.

Follow-up Treatment Subsequent follow-up would occur weekly for 4 weeks post inpatient treatment and then every 4 weeks to week 25. Patients will continue the same dose of Suvorexant/placebo for the duration of the follow-up period. At the end of the 25 week trial patients will continue to receive treatment as usual. If they wish to continue to receive suvorexant they can get a prescription from their GP (suvorexant has been added to the pharmaceutical benefits scheme).

Data Collection Baseline

* Name, date of birth, gender, contact details.
* ISI Insomnia Severity Index questionnaire (modified)
* Substance use history, medical history including current medications.
* Psychosocial status (data routinely collected through national minimum data set)
* Past history withdrawal symptoms ("delirium tremens", "seizures" etc)
* DSM 5 criteria for alcohol use disorder (AUD)
* Structured clinical Interview for DSm-5 (SCID-5)
* Pittsburgh Sleep Quality Index (PSQI)
* Epworth Sleepiness Scale
* K10 (Kessler Psychological Distress Scale), 10 questions about psychological distress symptoms: baseline and daily while in alcohol withdrawal then at monthly follow up
* ATOP Australian Treatment Outcome Profile
* Breath alcohol reading
* Liver function test
* Urine drug screen

In-patient withdrawal:

* Actigraphy measures of sleep patterns (Externally worn non-invasive accelerometer and light exposure recorder worn continually, from the first day of admission to discharge).
* Portable Polysomnography (Multichannel recoding of the electrophysiological markers of sleep). Polysomnography (PSG) records brain activity, eye movements and muscle tone to identify stages of sleep. In addition leg movements, heart rhythm, pulse rate, oxygen saturation, nasal breath flow, snore and chest movements are used to identify respiratory activity and lower leg muscle activity is also monitored for disturbing movements. (Day 1 and Day 7)
* Epworth Sleepiness Scale (excessive daytime sleepiness)
* Sleep diary during their stay (seven-ten days)
* ISI Insomnia questionnaire (Day 7 only)
* Clinical Information (as per open ended questioning for all AE's)
* CIWA-Ar (revised Clinical Institute Withdrawal Assessment for Alcohol scale), 10-item assessment of severity of alcohol withdrawal: baseline and every 2 - 4 hours, performed by trained staff
* Craving for alcohol using Obsessive Compulsive Drinking Scale
* Kessler 10 measure of psychological distress (Day 7 last 3 days)

At weekly follow-up, for weeks 2 to 5 and at monthly follow-up from week 9 to 25

* Pittsburgh Sleep Quality Index (sleep quality) (Wk5,9,13,17,21,25)
* Epworth Sleepiness Scale on admission (excessive daytime sleepiness)
* Sleep diary & ISI insomnia questionnaire
* Additional 2 short questions will be collected:

  * how many hours sleep has the participant had for the past week;
  * how would the participant rate their sleep quality in the past week;
* Clinical Information (as per open ended questioning for SAE safety data suvorexant form)
* Alcohol and other substance use (self report)
* ATOP Australian Treatment Outcome Profile (Wk5,9,13,17,21,25)
* K10 (Kessler Psychological Distress Scale)
* Breath alcohol reading
* Urine drug screen
* Liver/renal function tests (Wk 2,5,9,13,17,21,25)
* Craving for alcohol using Obsessive Compulsive Drinking Scale

Any differences between objective and subjective sleep measures will be documented and reflected back to patients on an individual basis. During the consent process all patients will be informed that this is a trial and that there will be no additional (other than the trial) medication provided for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and not more than 75 years of age
* DSM-5 diagnosis of insomnia
* Alcohol dependent (SCID-5)
* Willing to comply with treatment and follow-up requirements of study
* Able to give informed consent

Exclusion Criteria:

* Consumes less than 6 standard drinks per day.
* Not alcohol dependent (SCID-5)
* Unstable major psychiatric disorder e.g. active psychosis, significant PTSD.
* Currently taking medication having major interaction with suvorexant
* Pregnant (urine βHCG positive) or not using adequate contraception.
* Breast feeding.
* Severe hepatic impairment (Liver enzyme levels >five times normal level)
* Severe renal impairment (urine creatinine clearance < 30ml/h)
* Severe medical disorder e.g. epilepsy, cardiovascular disorder
* Participating in another pharmacotherapy trial e.g. lorcaserin
* Highly dependent on medical care.
* Driver of any vehicle (car or commercial vehicle)
* Inability to take oral medication.
* No consent to participate in the study
* Known sensitivity to suvorexant.
* Less than 18 years of age
* Over 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep measure | 7-10 days
  Change in polysomnography sleep efficiency measure from baseline and at end of inpatient stay. Portable Polysomnography is multichannel recording of the electrophysiological markers of sleep. Polysomnography (PSG) records brain activity, eye movements and muscle tone to identify stages of sleep. Sleep efficiency measure is number of minutes of sleep divided by the number of minutes in bed {%}).

SECONDARY OUTCOMES:
Sleep measure | 25 weeks
  Changed ISI scores from baseline at end of inpatient stay plus at 5 weeks, 9, 13, 17, 21, 25 weeks. The ISI is 7 questions (0-4) with a maximum score of 28 for severe insomnia. The investigators anticipate a change in total score.
Sleep quality: Pittsburgh Sleep Quality Index (PSQI) | 25 weeks
  Changed Pittsburgh Sleep Quality Index (PSQI) scores from baseline at end of inpatient stay plus at 5 weeks, 9, 13, 17, 21, 25 weeks. The PSQI is a battery of 9 questions (scores 0-3). A total score of 5 or more indicates poor sleep. The investigators anticipate a change in total score.
Sleepiness measure | 25 weeks
  Changed Epworth Sleepiness Scale scores from baseline at end of inpatient stay plus at 5 weeks, 9, 13, 17, 21, 25 weeks. There are 8 questions with scores of 0-3, maximum score of 24 indicates excessive sleepiness. A change in total score is anticipated.
Abstinence measure | 25 weeks
  Abstinence rates from baseline at 5 weeks, 9, 13, 17, 21, 25 weeks (%)
Relapse measure | 25 weeks
  Relapse to heavy drinking (>5 drinks/day) from baseline to 5 weeks, 9, 13, 17, 21, 25 weeks
Craving measure | 25 weeks
  Change in alcohol craving measures using the Obsessive Compulsive Drinking Scale from baseline at 5 weeks, 9, 13, 17, 21, 25 weeks. This scale is made up of 14 questions (0-4 range). The higher the total score, the greater the craving. The investigators anticipate a change in total score.
Liver function measure | 25 weeks
  Liver function change [Aspartate aminotransferase (AST) and Gamma-glutamyltransferase (GGT) levels] from baseline at 5 weeks, 9, 13, 17, 21, 25 weeks (%)
Urine drug screen | 25 weeks
  Urine drug screens negative for drugs other than alcohol from baseline at 5 weeks, 9, 13, 17, 21, 25 weeks (%)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lawrence, Principal Investigator — Florey Institute of Neuroscience & Mental Health; Yvonne Bonomo, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker LC, Lawrence AJ. The Role of Orexins/Hypocretins in Alcohol Use and Abuse. Curr Top Behav Neurosci. 2017;33:221-246. doi: 10.1007/7854_2016_55. PMID 27909991
- [Background] Lawrence AJ, Cowen MS, Yang HJ, Chen F, Oldfield B. The orexin system regulates alcohol-seeking in rats. Br J Pharmacol. 2006 Jul;148(6):752-9. doi: 10.1038/sj.bjp.0706789. Epub 2006 Jun 5. PMID 16751790
- [Background] von der Goltz C, Koopmann A, Dinter C, Richter A, Grosshans M, Fink T, Wiedemann K, Kiefer F. Involvement of orexin in the regulation of stress, depression and reward in alcohol dependence. Horm Behav. 2011 Nov;60(5):644-50. doi: 10.1016/j.yhbeh.2011.08.017. Epub 2011 Sep 16. PMID 21945150
- [Background] Brower KJ. Insomnia, alcoholism and relapse. Sleep Med Rev. 2003 Dec;7(6):523-39. doi: 10.1016/s1087-0792(03)90005-0. PMID 15018094
- [Background] Roehrs T, Roth T. Sleep, sleepiness, and alcohol use. Alcohol Res Health. 2001;25(2):101-9. PMID 11584549